CLINICAL TRIAL: NCT02594046
Title: The Effect of Allogeneic Human Adipose Derived Stem Cell Component Extract on Androgenic Alopecia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, professor, Pusan National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: L-2015-199-2
Record Dates: First submitted 2015-10-30; First posted 2015-11-02 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Androgenic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- stem cell group (Experimental): stem cell group who apply 1.2 g of allogeneic human adipose derived stem cell component extract on their scalp for 16 weeks
  Interventions: Other: stem cell component extract
- placebo group (Placebo Comparator): placebo group who apply a placebo on their scalp for 16 weeks
  Interventions: Other: stem cell component extract

INTERVENTIONS:
Other: stem cell component extract — The Allogeneic Human adipose derived stem cell component extract
  Other Names: Tiara hair toninc

SUMMARY:
This randomized, placebo-controlled, double-blind study evaluates the efficacy and tolerability of the allogeneic human adipose derived stem cell component extract on androgenic alopecia in relatively healthy adults. A total of 38 subjects received 1.2 g of allogeneic human adipose derived stem cell component extract per month or a placebo for 16 weeks.

DETAILED DESCRIPTION:
This randomized, placebo-controlled, double-blind study evaluates the efficacy and tolerability of the allogeneic human adipose derived stem cell component extract on androgenic alopecia in relatively healthy adults. A total of 38 subjects received 1.2 g of allogeneic human adipose derived stem cell component extract per month or a placebo for 16 weeks. Hair count and thickness will be primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* androgenic alopecia basic and specific(BASP) classification: M2, C2, U1, V1, or F1 or higher

Exclusion Criteria:

* patient of scalp disease

Ages: 19 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2015-07-01; Primary Completion 2016-02-28 (Actual); Study Completion 2016-05-28 (Actual)

PRIMARY OUTCOMES:
change of total hair counts by phototrichogram | 16 weeks

IPD SHARING:
Plan to Share IPD: No